CLINICAL TRIAL: NCT01150591
Title: The Role of Microaspiration in Idiopathic Pulmonary Fibrosis
Brief Title: Microaspiration in Pulmonary Fibrosis
Acronym: ROMI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: F32HL097383 (NIH)
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: This is a prospective cohort study of patients with IPF. Subjects will undergo (1) an assessment of the presence or absence of microaspiration (via bronchoscopy and BAL pepsin level), (2) measurement of biomarkers of microaspiration (via esophageal function studies, laboratory tests, pulmonary function, chest imaging, and survey), and (3) longitudinal follow-up to document disease progression (via pulmonary function and survey).
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis 1: Microaspiration, as diagnosed by bronchoalveolar lavage (BAL) pepsin, is common in patients with IPF.

Hypothesis 2a: Baseline clinical variables and co-morbid conditions are risk factors for microaspiration in patients with IPF.

Hypothesis 2b: Baseline biological variables reflecting alveolar epithelial injury and inflammation are markers of microaspiration in IPF.

Hypothesis 3a: Microaspiration will lead to a more rapid rate of decline in pulmonary function.

Hypothesis 3b: Microaspiration will lead to higher rates of urgent medical care use (i.e. unscheduled clinic visit, emergency room visit, or hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF
* Ability ot provide informed consent

Exclusion Criteria:

* History of fundoplication or other gastroesophageal surgery
* Too ill to undergo bronchoscopy in the opinion of the investigator

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPF
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
BAL pepsin level | Cross sectional

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Francisco, San Francisco, California, United States